CLINICAL TRIAL: NCT01237938
Title: Pilot Study of the Effect of a Low Glycemic Index Diet on Breast Density (Diet and Breast Health Study )
Brief Title: Effect of a Low Glycemic Index Diet on Breast Density
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: test
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 71005
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low Glycemic Diet (Experimental)
  Interventions: Behavioral: Low Glycemic Diet

INTERVENTIONS:
Behavioral: Low Glycemic Diet — Changing to low glycemic diet

SUMMARY:
This study is a Pilot Phase II cancer intervention trial of a low glycemic index diet to reduce mammographic density in women at high risk for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Are between 40 and 60 years of age
* Still menstruating with at least 10 menstrual cycles in the previous 12 months
* Not Taking hormone replacement therapy
* Stable oral contraceptive use (no changes is use in past 12 months nor changes intended during interventional period)
* Have not been previously diagnosed with breast cancer, DCIS,lobular carcinoma in situ, atypical lobular hyperplasia or atypical hyperplasia
* No history of breast augmentation or reduction surgery
* Have no history of any other malignancy (excluding non-melanoma skin cancer) in the previous 5 years
* Have no history of diabetes or other metabolic diseases requiring dietary modification
* Have a study baseline mammographic density of at least 50% as estimated by mammographer
* BIRADS 1 or 2 mammogram if first ever mammogram, otherwise stable mammogram (no change since previous year)
* Have not followed a weight reduction or Atkins typs diet in the past 6 months Not pregnant or lactating in the past 12 months, nor intending pregnancy during the study period
* Successful completion of three baseline telephone-administered 24- hour dietary recalls

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2006-03; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Diet Change | 2 years
  To Assess the feasibility of a randomized trial to achieve diet change and promote longterm adoption of a low glycemic index diet intervention among women at high risk for breast cancer (> 50% of breast area occupied by radiological density)

SECONDARY OUTCOMES:
Biomarkers | 4, 8 & 12 months on Treatment
  To estimate the effect of a low glycemic index diet on breast cancer related biomarkers, including those associated with carbohydrate, growth and steroid hormaone metabolism and mammograhic density. Result from this aim will provide important preliminary data for use in planning a larger clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Susan McCann, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States